CLINICAL TRIAL: NCT04399265
Title: A Randomised Controlled Trial on the Clinical Efficacy of Oral Trehalose in Patients With Spinocerebellar Ataxia 3: Clinical & FMRI Correlation
Brief Title: Efficacy Of Oral Trehalose In Spinocerebellar Ataxia 3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Dr Norlinah Mohamed Ibrahim, Professor, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DIP-2019-007
Record Dates: First submitted 2020-03-11; First posted 2020-05-22 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Spinocerebellar Ataxia Type 3
Keywords: Spinocerebellar ataxia Type 3; Cerebellar Cognitive and Affective Syndrome; Trehalose; Neuropsychology; Magnetic resonance imaging
MeSH Terms: conditions — Machado-Joseph Disease; Cerebellar Cognitive Affective Syndrome | interventions — Trehalose; Maltose

STUDY DESIGN:
Intervention Model Description: This study will employ a double-blind randomised controlled trial (RCT) with two arms. Patients with SCA3 will be randomly allocated to oral trehalose group and a maltose placebo group. A total of 20 participants will be allocated to each group. There is a possibility of including other types of SCA at later stage of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients with SCA 3 will be randomised into the active treatment group and placebo group to which they are blinded from their group allocation. Likewise, the outcome assessor will be blinded from the patient's group status. A partial unblinding will be made with Group A vs. Group B (rather than the actual grouping) for preliminary analysis on Visit 1 and Visit 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trehalose (Experimental): Trehalose powder form to be dissolved in water, to be consumed by mouth, every day for 3 months.
  Interventions: Dietary Supplement: Trehalose
- Maltose placebo (Placebo Comparator): Isocaloric maltose powder form to be dissolved in water, to be consumed by mouth, every day for 3 months.
  Interventions: Dietary Supplement: Maltose

INTERVENTIONS:
Dietary Supplement: Trehalose — A disaccharide sugar usually used as food preservative, but for this study it is given at a higher dose
  Arms: Trehalose
Dietary Supplement: Maltose — Maltose power
  Arms: Maltose placebo

SUMMARY:
This study evaluates the effectiveness of oral trehalose in alleviating the neuropathological and motor behaviour deficits among patients with SCA3. A total of 40 participants with SCA3 will be recruited, with 20 participants to be administered with trehalose while another 20 participants to be administered with a maltose placebo.

DETAILED DESCRIPTION:
Spinocerebellar ataxia 3 (SCA3) is a rare form of inherited neurodegenerative disease involving progressive degeneration of spinocerebellar tract. SCA3 is characterised by increasingly worsening cerebellar function leading to gait abnormalities and poor coordination, dysarthria, and abnormal eye movements. Non-ataxia features include pyramidal and extrapyramidal manifestations, sensorimotor, neuropsychological and psychiatric symptoms. This is attributed to the role of cerebellum in motor, cognitive and affective processing (i.e. cerebellar cognitive and affective syndrome; CCAS), as well as its extensive connection with cerebral structures.

Trehalose is an omnipotent disaccharide molecule found in lower and higher life forms except in vertebrates. It has an amorphous (i.e. non-reducing) property, which is shown in its high hydrophilicity, chemical stability and strong resistance to denaturation / breakdown by heat, acid or enzyme. It is also shown to help refold partially denatured protein, thereby stabilizes protein aggregates, including those of polyglutamine, in vivo as well as in vitro. This has provided an avenue in which trehalose as a therapeutic agent for neurodegenerative disorders with pathological changes of protein aggregates.

In this study, a double-blinded randomised controlled trial (RCT) will be employed. A total of 40 patients with SCA3 will be randomly allocated to oral trehalose group and a placebo group (20 participants for each arm). With regards to clinical outcomes, motor and cognitive performances will be assessed to infer the efficacy of trehalose. Likewise, structural, resting-state fMRI (i.e. functional connectivity), and MR spectroscopy (i.e. metabolism), will be used as imaging biomarkers in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years old.
* Genetically confirmed SCA 3 diagnosis.
* Presence of progressive cerebellar syndrome (i.e. symptomatic) and genetic confirmation of SCA 3 in one of the immediate family members with similar clinical syndrome.
* Able to read, speak, and understand English or Malay.

Exclusion Criteria:

* Diagnosis of Diabetes Mellitus Type 1 or Type 2
* Presence of any concomitant neurological condition that might interfere with clinical measures used in this study.
* Presence of contraindication or hypersensitivity to trehalose.
* Use of stimulant / medication, caffeine, and tobacco within less than 24 hours washout period prior to assessment and / or scan.
* Presence of severe visual and / or auditory perceptual deficits.
* MRI contra-indications: claustrophobia, pregnancy, electronic implants (e.g. pacemaker) in the body, aneurysm clip, and current or past employment as machinists, welders or metal workers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline Scale for Ataxia Rating Assessment (SARA) at 3 months, 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up. | Baseline, 3 months, and 6 months, as well as 3, 6, 9, and 12 months post-treatment follow-up.
  An 8-item scale to quantify the severity of ataxia with a scoring of 0 (no ataxia) to 40 (most severe ataxia). Total time taken for test administration is estimated at 10 minutes.

SECONDARY OUTCOMES:
Changes from Baseline Spinocerebellar Ataxia Functional Index (SCAFI) at 3 months and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up. | Baseline, 3 months, and 6 months, as well as 3, 6, 9, and 12 months post-treatment follow-up.
  A validated multi-modal assessment tool that is composed of: a) timed 8 metre walk (8MW); b) the 9-hole peg test (9HPT); and c) the rate of "PATA" repetition over 10 seconds (PATA) to rate speech performance. Total time taken for test administration is estimated at 10 minutes.
Changes from Baseline Inventory of Non-Ataxia Symptoms (INAS) at 3 months and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up. | Baseline, 3 months, and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up.
  A validated scale assessing non-cerebellar signs with a scoring of 0 (no non-ataxia sign) to 16 (all assessed systems affected). Total time taken for test administration is estimated at 10 minutes.
Changes from Baseline Cerebellar Cognitive & Affective Syndrome (CCAS) Scale at 3 months and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up. | Baseline, 3 months, and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up.
  CCAS Scale is a brief cognitive screening tool to help identify CCAS in patients with cerebellar impairment. It derives a total score of 120 as a continuous measure; as well as an ordinal measure in accordance to the number of failed tests: 1) Possible CCAS = 1 failed test; 2) Probable CCAS = 2 failed tests; Definite CCAS = 3 or more failed tests. Four different forms were available to minimize the practice effect. Total time taken for test administration is estimated at 10 minutes.
Changes from Baseline Wechsler Adult Intelligence Scale (WAIS - 4) at 3 months and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up. | Baseline, 3 months, and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up.
  WAIS - 4 is an IQ test designed to measure intelligence and cognitive ability in adults and older adolescents. The selected subtests are Matrix Reasoning, Digit Span, and Coding. These subtests are used to measure abstract reasoning, WM, and processing speed respectively. These index and subtests have good reliability
Changes from Baseline Delis-Kaplan Executive Function System (D - KEFS) at 3 months and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up. | Baseline, 3 months, and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up.
  D - KEFS is a neuropsychological battery designed to measure various subdomains of executive function from 8 - 89 years old. The selected subtests are: Tower Test, Trail Making Test (TMT), Colour-Word Interference Test (CWIT). These tests measure planning, set-shifting, and inhibition abilities respectively.
Changes from Baseline Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS Update) at 3 months and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up. | Baseline, 3 months, and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up.
  RBANS Update is a neuropsychological battery designed to measure 5 neuropsychological domains from 12:0 - 89:11 years old. The selected subtests are: Figure Copy and Figure Recall. These tests measure visual construction, visual memory, and language abilities respectively.
Changes from Baseline Resting state fMRI at 3 months. | Baseline and 3 months
  The level of measurement of oxy-Hb (activation level) is continuous; greater oxy-Hb (mM.mm) indicates greater activation.
Changes from Magnetic resonance spectroscopy at 3 months. | Baseline and 3 months
  The level of measurement of N-Acetyl Aspartate (NAA; metabolism) is continuous; greater NAA (ppm) indicates greater metabolism.

OTHER OUTCOMES:
Changes from Baseline Structural / T1 MRI at 3 months. | Baseline and 3 months
  The level of measurement of grey matter density (structural) is continuous; greater grey matter density indicates greater structural volume.
Changes from Baseline Situational Motivation Scale (SIMS) at 3 months and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up. | Baseline, 3 months, and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up.
  SIMS comprises 16 items on four subscales, Intrinsic motivation (e.g., "I think that this activity is interesting"), Identified regulation (e.g., "I am doing it for my own good"), External regulation (e.g., "I am supposed to do it") and Amotivation (e.g., "I don't see what this activity brings me"). It contains 4 items per subscale scored on a scale from 1 to 7 providing a score between 4 and 28 for each subscale. It has an internal reliability of α = .74 - .83 for the four subscales. Total time taken for test administration is estimated at 5 minutes.
Changes from Baseline EuroQol-5D 3L (EQ-5D-3L) at 3 months and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up. | Baseline, 3 months, and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up.
  EQ-5D-3L consists of 2 parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). EQ-5D has 5 dimensions of assessment (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 3 levels (ordinal): no problem, some problem, and extreme problem. It has an internal reliability of α = .83 and valid among clinically and demographically heterogeneous patients. Total time taken for test administration is estimated at 5 minutes.
Adverse event | Baseline, 3 months, and 6 months; as well as 3, 6, 9, and 12 months post-treatment follow-up.
  Adverse event will be recorded in terms of severity, study intervention relationship, action taken regarding study intervention, outcome of adverse event, expected, and serious adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Norlinah Mohamed Ibrahim, MRCP, Principal Investigator — National University of Malaysia
Locations (1):
- UKM Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No